CLINICAL TRIAL: NCT01943409
Title: Parenteral Nutrition in Hospitalized Patients: Comparison of Two Commercially Available Lipid Emulsions
Brief Title: Intravenous Nutrition in Hospitalized Patients: Comparison of Two Oils
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johane Allard (Other)
Responsible Party: Sponsor-Investigator, Johane Allard, Professor of Medicine, Director-Division of Gastroenterology, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CAPCR ID: 13-5807
Record Dates: First submitted 2013-07-17; First posted 2013-09-17 (Estimated); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Obstruction; Cancer; Ileus; Malnutrition; Surgery
Keywords: Parenteral nutrition; lipid emulsion; Intralipid; ClinOleic; Inflammation; Infection; Bloodstream Infection; length of stay; mortality
MeSH Terms: conditions — Bites and Stings; Neoplasms; Ileus; Malnutrition; Hyperphagia; Inflammation; Infections; Sepsis | interventions — soybean oil, phospholipid emulsion; ClinOleic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intralipid (Active Comparator): Patients will receive Intralipid, which is the standard lipid emulsion used in the hospital
  Interventions: Drug: Intralipid
- ClinOleic (Experimental): Patients that are randomized to receive ClinOleic as a lipid emulsion in their PN, instead of Intralipid. ClinOleic is approved by Health Canada. The amount of calories from the lipid emulsion will be equivalent in the standard of care group and in the ClinOleic group.
  Interventions: Drug: ClinOleic

INTERVENTIONS:
Drug: Intralipid — soybean oil-based lipid emulsion
  Arms: Intralipid
Drug: ClinOleic — olive oil-based lipid emulsion
  Arms: ClinOleic

SUMMARY:
Intravenous nutrition is an important therapy for the recovery of many patients. It is indicated when the patients cannot take food by mouth or use their intestines for feeding. It is important to indicate it in the appropriate setting because it's not free of complications and is a costly treatment. Some of the complications are: elevated blood sugar or lipids, elevated liver function tests, infection of the catheter or device used to administer intravenous nutrition. Intravenous nutrition is composed by proteins, lipids, carbohydrates (sugar in the form of glucose) and vitamins. Until recently, Intralipid, a soybean oil-based lipid emulsion was the only lipid available in Canada for this kind of nutrition. Since 2010, a new lipid emulsion (ClinOleic) based on olive-oil has been approved by Health Canada for use in intravenous nutrition. There is an increasing need for hospitals to evaluate the quality of intravenous nutrition administered to hospitalized patients in terms of: assessing indications, prescription, complications, clinical results and costs. The objective of this study is to determine if intravenous nutrition prescribed in hospitalized patients is indicated following existing guidelines in terms of timing of nutrition support, prescription, monitoring and whether it is associated with complications. In addition, length of stay and mortality will be assessed. Also, we will evaluate nutritional, infectious and inflammatory parameters in patients receiving soybean oil-based lipid emulsion (Intralipid) compared to those of patients receiving olive oil-based lipid emulsion (ClinOleic).

DETAILED DESCRIPTION:
Until recently, Intralipid, a soybean oil-based lipid emulsion, has been the only available lipid for intravenous use in Canada. In 2010, ClinOleic, a new, predominantly olive oil based emulsion, has been approved by Health Canada as an alternative lipid.

There is an increasing need for hospitals to do quality-assurance studies for in-patient parenteral nutrition (PN) to assess indications, PN prescription, complications, clinical outcomes and costs. The only in-patient population that is well studied is the intensive care unit (ICU) population. Several meta-analyses showed that PN was associated with higher infection rate, longer length of stay and higher mortality when compared with enteral nutrition. Results from these and other studies were the basis for the Canadian ICU Guidelines.

The aim of this study is to determine if PN prescribed in in-patients is indicated, appropriately following existing guidelines in terms of timing of nutrition support, prescription and monitoring and, whether it is associated with complications. In addition, clinical outcomes such as length of stay and mortality will be assessed. Also, we will evaluate metabolic, nutritional, infectious and inflammatory parameters in patients receiving soybean oil-based lipid emulsion compared to those of patients receiving olive oil-based lipid emulsion.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older

  * Patients with PN during their hospitalization
  * Patients hospitalized in medical, surgical or ICU wards
  * Signed informed consent either from the patient, their legally authorized representative or a direct family member

Exclusion Criteria:

* • Patients without PN during their hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johane P Allard, MD, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intralipid | ClinOleic
Started | 153 | 150
Completed | 108 | 102
Not Completed | 45 | 48
Not completed — resumed oral/entral | 24 | 20
Not completed — Protocol Violation | 14 | 24
Not completed — Death | 3 | 1
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Baseline Characteristics: Baseline Characteristics between Clinoleic and Intralipid
Arm/Group | Baseline Characteristics
Number analyzed (Participants) | 210
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: These are the baseline characteristics compared between groups
  years
    ClinOleic: number analyzed (Participants) | 102
    ClinOleic | 56.81 (14.06)
    Intralipid: number analyzed (Participants) | 108
    Intralipid | 57.18 (16.43)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: This is the comparison between groups
  Participants
    ClinOleic: number analyzed (Participants) | 102
    ClinOleic: Female | 53
    ClinOleic: Male | 49
    Intralipid: number analyzed (Participants) | 108
    Intralipid: Female | 68
    Intralipid: Male | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Pre-albumin [Mean (Standard Deviation); unit: g/l] — Population: comparison between groups
  g/l
    Clinoleic: number analyzed (Participants) | 102
    Clinoleic | 0.10 (0.15)
    Intralipid: number analyzed (Participants) | 108
    Intralipid | 0.11 (0.16)

OUTCOME MEASURES:

1. Primary Outcome: Prealbumin
Description: prealbumin is an hepatic protein that is used in the diagnosis of malnutrition. It has a short half-life so any changes in nutritional status can rapidly be represented by prealbumin levels.
Time Frame: at day 10
Measure: Mean (Standard Deviation); unit: g/l
Arm/Group | Intralipid | ClinOleic
Number analyzed (Participants) | 108 | 102
g/l | 0.15 (0.08) | 0.16 (0.08)

2. Secondary Outcome: Length of Stay
Description: Length of stay in the hospital and ICU will be recorded for 1 year
Time Frame: participants will be followed for the duration of hospital stay up to one year
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intralipid | ClinOleic
Number analyzed (Participants) | 108 | 102
days | 45.63 (41.45) | 40.18 (36.60)

3. Secondary Outcome: Mortality
Description: We will follow the patients from the day of admission until the day of discharge and record the mortality for 1 year
Time Frame: participantes will be followed for the duration of hospital stay for up to 1 year
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intralipid | ClinOleic
Number analyzed (Participants) | 108 | 102
days | 11 (10.19) | 13 (12.75)

4. Secondary Outcome: Infections
Description: we will record the infections the patients develop during PN until one week after PN for 1 year
Time Frame: until one week post-PN up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Intralipid | ClinOleic
Number analyzed (Participants) | 108 | 102
Participants | 36 | 40

5. Secondary Outcome: Change in Hand-grip Strength
Description: We will measure hand grip strength at baseline (day0) and at day 10 of PN. This is a test that measures the strength of the hand and forearm muscles and is often used as a general test of strength
Time Frame: at baseline (day 0) and day 10 of PN
Measure: Mean (Standard Deviation); unit: Kilogram
Arm/Group | Intralipid | ClinOleic
Number analyzed (Participants) | 108 | 102
Kilogram | 0.10 (4.97) | -0.35 (4.70)

6. Secondary Outcome: Change in Mid-arm Circumference
Description: This is a rough indicator of body fat
Time Frame: at baseline (day0) and day 10
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intralipid | ClinOleic
Number analyzed (Participants) | 108 | 102
cm | -0.27 (1.04) | -0.18 (1.67)

7. Secondary Outcome: Subjective Global Assessment (SGA): Number Who Improved
Description: is a bedside method that assesses the risk of malnutrition and identifies which patient will benefit best from nutrition support
Time Frame: at baseline (day 0) and day 10
Measure: Count of Participants; unit: Participants
Arm/Group | Intralipid | ClinOleic
Number analyzed (Participants) | 108 | 102
Participants | 12 | 15

8. Secondary Outcome: Change in High Sensitivity C-reactive Protein (Hs-CRP)
Description: hs-CRP is a marker of inflammation, we will measure this parameter at baseline and after 10 days of PN
Time Frame: Baseline (day 0) and day 10
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Intralipid | ClinOleic
Number analyzed (Participants) | 108 | 102
mg/dl | -23.52 (79.99) | -29.42 (70.47)

9. Secondary Outcome: Red Blood Cell Fatty Acid Composition: Linoleic
Description: Red blood cell fatty acid composition, particularly the essential fatty acids (linoleic acid and alpha-linolenic acid) will be measured to assess presence/absence of essential fatty acid deficiency
Time Frame: day 10
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Intralipid | ClinOleic
Number analyzed (Participants) | 108 | 102
ug/ml | 578.34 (315.40) | 845.96 (365.58)

ADVERSE EVENTS:
Time Frame: Through study completion up to 1 year
Arm/Group | Intralipid | ClinOleic
All-Cause Mortality (participants affected / at risk) | 3/153 | 1/150
Serious Adverse Events (participants affected / at risk) | 0/153 | 1/150
Other Adverse Events (participants affected / at risk) | 0/153 | 0/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intralipid (N=153) | ClinOleic (N=150)
Line infection (Infections and infestations) | NA | 1 (1) — Patient was removed from study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-13): https://cdn.clinicaltrials.gov/large-docs/09/NCT01943409/Prot_SAP_001.pdf